CLINICAL TRIAL: NCT00043134
Title: Intravenous Low-Dose Decitabine Versus Supportive Care in Elderly Patients With Primary Myelodysplastic Syndrome (MDS) (>10% Blasts or High-Risk Cytogenetics), Secondary MDS or Chronic Myelomonocytic Leukemia (CMML) Who Are Not Eligible for Intensive Therapy: An EORTC-German MDS Study Group Randomized Phase III Study
Brief Title: Low-Dose Decitabine Compared With Standard Supportive Care in Treating Older Patients With Myelodysplastic Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000256224; EORTC-06011; SUPERGEN-EORTC-06011; GMDSG-EORTC-06011; EudraCT-2005-002830
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2008-04

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; refractory anemia; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; refractory anemia with ringed sideroblasts; refractory cytopenia with multilineage dysplasia; secondary myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myelomonocytic, Chronic; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders | interventions — Decitabine

INTERVENTIONS:
Drug: decitabine

SUMMARY:
RATIONALE: Decitabine may help myelodysplasia cells develop into normal stem cells. It is not yet known if decitabine is more effective than standard supportive care in treating myelodysplastic syndrome.

PURPOSE: Randomized phase III trial to compare the effectiveness of low-dose decitabine with that of standard supportive care in treating older patients who have myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of low-dose decitabine vs standard supportive care, in terms of overall survival, of elderly patients with myelodysplastic syndromes.
* Compare the response rate and progression-free survival of patients treated with these regimens.
* Determine the toxicity of decitabine in these patients.
* Assess the duration of hospitalization and number of blood transfusions in patients treated with these regimens.
* Assess the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to cytogenetic risk factors (good vs poor vs intermediate vs unknown), disease (primary myelodysplastic syndrome (MDS) vs secondary MDS), and participating center. Patients with a successful cytogenetic exam are also stratified according to overall International Prognostic Scoring System score (intermediate 1 vs intermediate 2 vs high risk). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive decitabine IV over 4 hours every 8 hours for 3 days. Treatment repeats every 6 weeks for 4-8 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive standard supportive care. Quality of life is assessed at baseline, every 6 weeks during therapy, every 2 months for 1 year, and then every 3 months thereafter.

Patients are followed every 2 months for 1 year and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 220 patients (110 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary or secondary myelodysplastic syndromes (MDS)

  * Any FAB or WHO criteria cellular type allowed
* Bone marrow blast count on aspiration or biopsy of 1 of the following:

  * No more than 10% with poor cytogenetic risk factors (defined as any numerical or structural abnormality of chromosome 7 and/or complex abnormalities)
  * 11-20%
  * 21-30% for patients with acute myeloid leukemia (AML) secondary to MDS (i.e., refractory anemia with excess blasts in transformation by FAB classification)
  * Patients who failed the cytogenetic exam are allowed provided bone marrow blasts are at least 5% and/or 2-3 cytopenias are present
* No rapid progression towards full-blown AML
* No blast crisis of chronic myeloid leukemia
* No t(8;21) alone or in combination with other abnormalities
* Ineligible for intensive chemotherapy (e.g., cytarabine or an anthracycline)

PATIENT CHARACTERISTICS:

Age

* 60 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* Hepatitis B surface antigen negative

Renal

* Creatinine less than 1.5 times ULN

Cardiovascular

* No severe cardiovascular disease
* No arrhythmias requiring chronic treatment
* No congestive heart failure
* No New York Heart Association class III or IV heart disease
* No symptomatic ischemic heart disease

Other

* HIV negative
* No active uncontrolled infection
* No other malignancy within the past 3 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix within the past 2 years
* No prior or concurrent evidence of CNS or psychiatric disorders requiring hospitalization
* No psychological, familial, sociological, or geographical condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 6 weeks since prior growth factors for primary MDS
* No concurrent antiangiogenic drugs (e.g., thalidomide)
* No concurrent interleukin, interferon, or anti-thymocyte globulin

Chemotherapy

* See Disease Characteristics
* More than 6 weeks since prior hydroxyurea for primary MDS
* No other prior chemotherapy for MDS or AML
* Prior chemotherapy for solid tumors or lymphoma (resulting in secondary MDS) allowed

Endocrine therapy

* No concurrent steroids (except as inhalation therapy)

Radiotherapy

* Prior radiotherapy for solid tumors or lymphoma (resulting in secondary MDS) allowed

Surgery

* Not specified

Other

* More than 6 weeks since prior immunosuppressive agents for primary MDS
* No concurrent amifostine
* No concurrent cyclosporine
* No other concurrent experimental therapies

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2002-05; Primary Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
Duration of overall survival

SECONDARY OUTCOMES:
Best response rate as measured by Cheson response criteria
Overall progression-free survival
Toxicity as assessed by CTC v2.0
Quality of life as assessed by EORTC QLQ30
Days in Hospital

CONTACTS AND LOCATIONS:
Overall Officials: Pierre W. Wijermans, MD, PhD — HagaZiekenhuis - Locatie Leyenburg; Michael Luebbert, MD — University Hospital Freiburg
Locations (46):
- Austria (2):
  - Innsbruck Universitaetsklinik, Innsbruck
  - St. Johanns-Spital, Salzburg
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - U.Z. Gasthuisberg, Leuven
  - H. Hartziekenhuis - Roeselaere., Roeselare
  - Centre Hospitalier Peltzer-La Tourelle, Verviers
- University Hospital Rebro, Zagreb, Croatia
- Czechia (2):
  - First Medical Clinic of Charles University Hospital, Prague
  - Institute of Hematology and Blood Transfusion, Prague
- Germany (24):
  - Charite University Hospital - Campus Virchow Klinikum, Berlin
  - Staedtisches Klinikum Braunschweig, Braunschweig
  - DIAKO Ev. Diakonie Krankenhaus gGmbH, Bremen
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - St. Johannes Hospital - Medical Klinik II, Duisburg
  - St. Antonius Hospital, Eschweiler
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Klinikum der Albert - Ludwigs - Universitaet Freiburg, Freiburg im Breisgau
  - Klinik Fuer Innere Medizin, Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - Medizinische Hochschule Hannover, Hanover
  - Ruprecht - Karls - Universitaet Heidelberg, Heidelberg
  - Universitaetsklinikum des Saarlandes, Homburg
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Onkologische Schwerpunktpraxis - Leer, Leer
  - Sana Kliniken Luebeck, Lübeck
  - Kreiskrankenhaus Luedenscheid, Lüdenscheid
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Staedtisches Krankenhaus Muenchen - Harlaching, Munich
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Southwest German Cancer Center at Eberhard-Karls-University, Tübingen
  - Klinikum Der Stadt Villingen - Schwenningen, Villingen-Schwenningen
  - Medizinische Poliklinik, Universitaet Wuerzburg, Würzburg
- Italy (5):
  - Universita Degli Studi di Florence - Policlinico di Careggi, Florence
  - Azienda Ospedaliera Vito Fazzi, Lecce
  - Azienda Ospedale - d S. Salvatore, Pesaro
  - Istituto Regina Elena, Rome
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
- Netherlands (5):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Leiden University Medical Center, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - HagaZiekenhuis - Locatie Leyenburg, The Hague
- Kantonsspital - Abteilung Onkologie, Basel, Switzerland
- Ibn-i Sina Hospital, Ankara, Turkey (Türkiye)
- Royal South Hants Hospital, Southampton, England, United Kingdom

REFERENCES:
- [Result] WijerMans P, Suciu S, Baila L, et al.: Low dose decitabine versus best supportive sare in elderly patients with intermediate or high risk MDS not eligible for intensive chemotherapy: final results of the randomizedpPhase III study (06011) of the EORTC Leukemia and German MDS Study Groups. [Abstract] Blood 112 (11): A-226, 2008.